CLINICAL TRIAL: NCT04959071
Title: Comparison of the Mean Healing Time of Wound After Vacuum Assisted Closure (VAC) Versus Conventional Dressing in Diabetic Foot Ulcer Patients
Brief Title: Mean Healing Time of Wound After Vacuum Assisted Closure (VAC) Versus Conventional Dressing in Diabetic Foot Ulcer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Mehwish Mooghal , MBBS, Resident Surgery at PNS Shifa Hospital Karachi, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAC vs Conventional Dressing
Record Dates: First submitted 2021-06-25; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Foot Ulcer; Healing Delayed; Wound; Foot; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Foot; Foot Injuries; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized control trial. After informed, written consent, all selected cases were offered to pick up a slip from total mixed up slips (half-slips contained letter 'A' and other half slips contained letter 'B') and he/she was placed in that respective group. In group A patients, VAC dressing was applied while in group B conventional dressing was applied. All patients were followed regularly by the single researcher and mean healing time was noted in every patient of both groups . This all data (age, gender, duration of ulcer, and size of ulcer, BMI, and healing time) was recorded on a specially designed Performa designed beforehand.
Who Masked: Participant
Masking Description: After informed, written consent, all selected cases were offered to pick up a slip from total mixed up slips (half-slips contained letter 'A' and other half slips contained letter 'B') and he/she was placed in that respective group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Group A included participants who underwent VAC therapy for diabetic Foot ulcers
  Interventions: Procedure: Vacuum assisted closure VAC vs conventional dressing
- Group B (Active Comparator): Group B included participants who underwent conventional dressings for diabetic foot ulcers
  Interventions: Procedure: Vacuum assisted closure VAC vs conventional dressing

INTERVENTIONS:
Procedure: Vacuum assisted closure VAC vs conventional dressing — In participants undergoing vacuum assisted closure a drainage tube was placed in the wound followed by dressing with sterile foam sheet and application of occlusive transparent film over the whole assembly. The drainage tube was connected to a suction machine. Intermittent negative pressure of -125mmHg was applied every 15 minutes; the suction was stopped for 10 minutes. The dressing was changed every 48 hours.
  In participants with conventional dressings, after wound wash, pyodine soaked gauze pieces were used for initial 48 hours followed by dressings of normal saline soaked gauze pieces, twice daily.
  Other Names: Conventional Dressing

SUMMARY:
Comparison the mean healing time of wound after vacuum assisted closure(VAC) versus conventional dressing(CD) in diabetic foot ulcer(DFU) patients.

DFUs are chronic wounds in diabetics resulting from ischemia, angiogenesis defects and impaired immunity. Different treatment modalities are available for treating DFUs. Amongst them VAC provides a new paradigm for diabetic wound dressing. Different studies concluded that DFUs treated with VAC are more likely to heal than CD.

The average healing time varies greatly among different studies conducted. Therefore, we conducted this study to compare the mean healing time of wound after VAC and CD in DFU patients. Based on these results, the method with lesser healing time can be opted for our routine practice guidelines for DFU patient's management protocol.

DETAILED DESCRIPTION:
This Randomized controlled trial was conducted at Department of General Surgery, at a tertiary teaching hospital , over duration of six months from 28th February 2020 to 27th August 2020. The calculated sample size was 60 i.e. 30 cases in each group, with 5% level of significance, 80% power of study and taking mean healing time with VAC therapy as 11.366 ± 3.488 days and with conventional dressing as 16.41 ± 3.104 days.6 Non-probability, consecutive sampling technique was used.

After taking permission from ethical review committee , total 60 patients who were presented in outpatient Department of Surgery, at a tertiary care Hospital, Karachi, fulfilling the inclusion criteria was selected. After informed, written consent, all selected cases were offered to pick up a slip from total mixed up slips (half-slips contained letter 'A' and other half slips contained letter 'B') and he/she was placed in that respective group. In group A patients, VAC dressing was applied while in group B conventional dressing was applied. In patients undergoing vacuum assisted closure a drainage tube was placed in the wound followed by dressing with sterile foam sheet and application of occlusive transparent film over the whole assembly. The drainage tube was connected to a suction machine. Intermittent negative pressure of -125mmHg was applied every 15 minutes; the suction was stopped for 10 minutes. The dressing was changed every 48 hours. In patients with conventional dressings, after wound wash, pyodine soaked gauze pieces were used for initial 48 hours followed by dressings of normal saline soaked gauze pieces, twice daily. All patients were followed regularly by the single researcher and mean healing time was noted in every patient of both groups as described in operational definition. This all data (age, gender, duration of ulcer, and size of ulcer, BMI, and healing time) was recorded on a specially designed Performa designed beforehand.

ELIGIBILITY:
Inclusion Criteria:

1. All patients with diabetic foot ulcer of >2 weeks duration. 2. Size of ulcer >3 cm. 3. Well controlled diabetes (HbA1C=6-8.3%). 4. Age 25-65 years. 5. Both genders.

-

Exclusion Criteria:

1. Anemic patients (hemoglobin <10 g/dl).
2. Patients with history of steroid intake.
3. Patients with chronic renal failure (assessed on history and s/creatinine >1.5 mg/dl).
4. Patients with history of immunosuppressive therapy.
5. Ulcers involving bone as well.

   -

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Comparison of mean healing time of wounds in diabetic foot ulcers among Vac and conventional dressings | 1 month
  participants were assessed for mean healing time of wound after VAC theray and conventional dressing. All participants were followed regularly by the single researcher and mean healing time was noted in every patient of both groups . Healing time was measured in number of days. The start time was the application of first VAC and end time will be the day of wound healing (appearance of granulation tissue over wound as assessed clinically). Similarly start time in conventional dressings was from day of first application of conventional dressing till appearance of granulation tissues over the wound. In both groups mean healing time was compared to see any difference in healing time of both the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University Medical and Dental College Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lone AM, Zaroo MI, Laway BA, Pala NA, Bashir SA, Rasool A. Vacuum-assisted closure versus conventional dressings in the management of diabetic foot ulcers: a prospective case-control study. Diabet Foot Ankle. 2014 Apr 8;5. doi: 10.3402/dfa.v5.23345. eCollection 2014. PMID 24765245
- [Background] Ravari H, Modaghegh MH, Kazemzadeh GH, Johari HG, Vatanchi AM, Sangaki A, Shahrodi MV. Comparision of vacuum-asisted closure and moist wound dressing in the treatment of diabetic foot ulcers. J Cutan Aesthet Surg. 2013 Jan;6(1):17-20. doi: 10.4103/0974-2077.110091. PMID 23723599
- [Background] Lavery LA, Murdoch DP, Kim PJ, Fontaine JL, Thakral G, Davis KE. Negative Pressure Wound Therapy With Low Pressure and Gauze Dressings to Treat Diabetic Foot Wounds. J Diabetes Sci Technol. 2014 Mar;8(2):346-349. doi: 10.1177/1932296813519012. Epub 2014 Feb 18. PMID 24876586
- [Background] James SMD, Sureshkumar S, Elamurugan TP, Debasis N, Vijayakumar C, Palanivel C. Comparison of Vacuum-Assisted Closure Therapy and Conventional Dressing on Wound Healing in Patients with Diabetic Foot Ulcer: A Randomized Controlled Trial. Niger J Surg. 2019 Jan-Jun;25(1):14-20. doi: 10.4103/njs.NJS_14_18. PMID 31007506